CLINICAL TRIAL: NCT00415805
Title: A Pilot, Open-label, Multicenter Intra-individual Comparison of Multihance and Vasovist for Contrast-Enhanced Magnetic Resonance Angiography (CE-MRA) of Renal Arteries
Brief Title: Renal MRA Crossover Study Comparing Multihance to Another Contrast Agent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: MH 128
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2009-03

CONDITIONS: Steno-occlusive Disease
MeSH Terms: interventions — gadobenic acid; gadofosveset trisodium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Multihance
- 2 (Active Comparator)
  Interventions: Drug: vasovist

INTERVENTIONS:
Drug: Multihance — 0.5 Molar, single injection at 0.2 mL/kg
  Arms: 1
Drug: vasovist — 0.25 molar single injection 0.03 ml/kg
  Arms: 2

SUMMARY:
This is an explorative small pilot study comparing two MRA contrast agents, one of which has been on the market for a few years and the other fairly new to the market. Since the study is explorative and designed to provide preliminary information for consideration for a future larger study, sample size is not based on statistical assumptions.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected renovascular disease based on one of the following criteria:

  * severe hypertension
  * hypertension refractory to standard therapy
  * abrupt onset of moderate to severe hypertension at age < 35 years
  * normalized blood pressure by an ACE inhibitor in a patient with moderate or severe hypertension
  * unexplained by stable elevation of serum creatinine > 2Mg/dL
  * positive findings for stenosis from another imaging modality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity compared to DSA | post dose

SECONDARY OUTCOMES:
accuracy and predictive values; inter-reader agreement for diagnostic performance | post dose

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics
Locations (1):
- Bracco Imaging, S.p.A, Milan, Italy